CLINICAL TRIAL: NCT02573961
Title: Laser Acupuncture Versus High Protein/Low Carbohydrate Diet on Endothelial Markers in Obese Females. A Randomized Controlled Trial
Brief Title: Laser Acupuncture Versus High Protein/Low Carbohydrate Diet on Endothelial Markers in Obese Females
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This was a topic for a thesis project where the topic was changed
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRCEgypt
Record Dates: First submitted 2015-10-05; First posted 2015-10-12 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2015-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, High-Protein Low-Carbohydrate; Caloric Restriction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- laser (Active Comparator): Subjects will receive 24 activated laser acupuncture group treatments. The laser will be applied for 10 seconds to each of the selected acupuncture points. In addition they will be instructed to take a tailored low caloric diet
  Interventions: Device: Laser acupuncture; Behavioral: low caloric diet
- high protein low carbohydrate diet (Active Comparator): Subjects will be instructed to take a tailored high protein/low carbohydrate/low caloric diet.
  Interventions: Behavioral: high protein low carbohydrate diet
- control (Sham Comparator): Subjects in the control group will undergo sham laser acupuncture treatment with no laser power output. In addition they will be instructed to take a tailored low caloric diet .
  Interventions: Device: Laser acupuncture; Behavioral: low caloric diet

INTERVENTIONS:
Device: Laser acupuncture — GaAlAs semiconductor diode Laser Phototherapy Device
  Arms: control; laser
Behavioral: high protein low carbohydrate diet — A tailored high protein/low carbohydrate/low caloric diet
  Arms: high protein low carbohydrate diet
Behavioral: low caloric diet — Tailored balanced low caloric diet
  Arms: control; laser

SUMMARY:
The purpose of this study is to compare the effects of laser acupuncture and high protein low carbohydrate diet on the treatment of obesity and lowering of endothelial markers.

DETAILED DESCRIPTION:
Sixty females above 20 years of age with a body mass index (BMI) of over 30 kg/m2 will be divided into three groups (20 in each): two experimental groups (laser; high protein low carbohydrate diet) and control. Each subject will receive the treatment relevant to their group, in addition to obtaining 3 days dietary recalls and measurements including BMI, serum insulin and endothelial markers. Laser and control group will receive 24 activated or sham laser acupuncture treatments. High protein low carbohydrate group will be instructed to take a tailored high protein/low carbohydrate diet.

ELIGIBILITY:
Inclusion Criteria:

* obese females of BMI more than 30 kg/m2, and
* of age range from 20 to 50 years.

Exclusion Criteria:

* medical history of chronic diseases,
* pregnancy,
* photosensitivity reactions to laser treatment,
* a pacemaker,
* medications known to affect one's weight up to 1 month in advance, or
* are unwilling to comply with the study protocol.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
weight loss | 8 weeks

SECONDARY OUTCOMES:
decrease cardiovascular risks | 8 weeks
  endothelial markers , serum insulin and insulin resistance changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Neveen H Abou El-Soud, Ph.D, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Ziccardi P, Nappo F, Giugliano G, Esposito K, Marfella R, Cioffi M, D'Andrea F, Molinari AM, Giugliano D. Reduction of inflammatory cytokine concentrations and improvement of endothelial functions in obese women after weight loss over one year. Circulation. 2002 Feb 19;105(7):804-9. doi: 10.1161/hc0702.104279. PMID 11854119
- [Background] Soenen S, Bonomi AG, Lemmens SG, Scholte J, Thijssen MA, van Berkum F, Westerterp-Plantenga MS. Relatively high-protein or 'low-carb' energy-restricted diets for body weight loss and body weight maintenance? Physiol Behav. 2012 Oct 10;107(3):374-80. doi: 10.1016/j.physbeh.2012.08.004. Epub 2012 Aug 19. PMID 22935440